CLINICAL TRIAL: NCT02005380
Title: Usability Study of Spaced Retrieval Exercise Using Mobile Devices for Alzheimer's Disease Rehabilitation
Status: Completed | Type: Observational
Sponsor: German-Jordanian University (Other)
Responsible Party: Principal Investigator, Ahmad Zmily, Assistant Professor, German-Jordanian University
Other Study IDs: GJU001
Record Dates: First submitted 2013-11-29; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease Rehabilitation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Text-based Task: This group is required to do the text-based task
  Interventions: Other: Text-based task
- Graphic-based Task: This group is required to do the graphic-based task
  Interventions: Other: Graphic-based Task

INTERVENTIONS:
Other: Text-based task — Participants are required to take text-based exercise.
  Groups: Text-based Task
Other: Graphic-based Task — Participants are required to take the graphic-based exercise.
  Groups: Graphic-based Task

SUMMARY:
The focus of this work is to explore the use of modern mobile technology to enable people with Alzheimer's disease to improve their abilities to perform activities of daily living and hence to promote independence and participation in social activities. This work also aims at reducing the burden on caregivers by increasing the AD patients' sense of competence and ability to handle behavior problems.

DETAILED DESCRIPTION:
The investigators developed ADcope, an integrated application that includes several modules that target individuals with Alzheimer's disease , using mobile devices. The investigators developed two different user interfaces: a text-based and a graphic-based. To evaluate the usability of the application, participants with early stages of AD were asked to run the two user interfaces of the spaced retrieval memory exercise using a tablet mobile device.

ELIGIBILITY:
Inclusion Criteria:

- Have early stages of Alzheimer's decease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Darat Samir Shamma, a senior residential care facility and
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
NASA Task Load Index Measure | 1 hour
  NASA-TLX is a multi-dimensional rating procedure that derives an overall workload score based on a weighted average of ratings on six subscales. These subscales include Mental Demands, Physical Demands, Temporal Demands, Own Performance, Effort, and Frustration.

SECONDARY OUTCOMES:
Test Score | 1 Hour
  Test score measures the percentage of questions answered by the participants correctly from the first trial.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Zmily, PhD, Principal Investigator — German-Jordanian University
Locations (1):
- Darat Samir Shamma, Amman, Amman Governorate, Jordan